CLINICAL TRIAL: NCT06985277
Title: Diagnostic Yield of Urgent Panendoscopy VS. Conventional Endoscopic Evaluation in Patients Presenting With Hematochezia : Randomized Controlled Trial
Brief Title: Urgent Panendoscopy in Patients Presenting With Hematochezia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nonthalee Pausawasdi, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Si265/2024
Record Dates: First submitted 2025-05-01; First posted 2025-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Lower Gastrointestinal Bleeding; Small Bowel Bleeding
Keywords: Hematochezia; colonoscopy; video capsule endoscopy; diagnostic yield
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Urgent colonoscopy with urgent VCE group (Experimental): Intervention Arm : Urgent colonoscopy with urgent VCE group :
  Patients will undergo colonoscopy within 24 hours of diagnosed lower gastrointestinal bleeding. If no bleeding source is identified on colonoscopy or presumed diverticular bleeding cases, esophagogastroduodenoscopy (EGD) followed by same-session video capsule endoscopy (VCE) will be performed immediately
  Interventions: Diagnostic Test: Urgent endoscopy strategy
- Standard colonoscopy with standard VCE group (Experimental): Control Arm : Standard colonoscopy with standard VCE group :
  Patients will undergo colonoscopy within 24-48 hours after diagnosed lower gastrointestinal bleeding. If no bleeding source is identified on colonoscopy or presumed diverticular bleeding cases, esophagogastroduodenoscopy (EGD) will be performed immediately. If EGD shows no bleeding source, video capsule endoscopy (VCE) will be performed within 24 hours of the preceding endoscopies
  Interventions: Diagnostic Test: Standard colonoscopy with standard VCE group

INTERVENTIONS:
Diagnostic Test: Urgent endoscopy strategy — Patients will undergo colonoscopy within 24 hours of diagnosed lower gastrointestinal bleeding. If no bleeding source is identified on colonoscopy or presumed diverticular bleeding cases, esophagogastroduodenoscopy (EGD) followed by same-session video capsule endoscopy (VCE) will be performed immediately
  Arms: Urgent colonoscopy with urgent VCE group
Diagnostic Test: Standard colonoscopy with standard VCE group — Patients will undergo colonoscopy within 24-48 hours after diagnosed lower gastrointestinal bleeding. If no bleeding source is identified on colonoscopy or presumed diverticular bleeding cases, esophagogastroduodenoscopy (EGD) will be performed immediately. If EGD shows no bleeding source, video capsule endoscopy (VCE) will be performed within 24 hours of the preceding endoscopies
  Arms: Standard colonoscopy with standard VCE group

SUMMARY:
Gastrointestinal bleeding is a significant emergency condition requiring prompt diagnosis. Current evidence presents a clinical paradox: urgent colonoscopy (within 24 hours) shows no clear benefit in several studies, while urgent video capsule endoscopy (VCE) demonstrates improved detection rates for small bowel bleeding.

This study aims to evaluate a novel approach combining urgent colonoscopy followed by same-day VCE for patients with normal colonoscopy findings. This strategy has not been previously assessed and may improve bleeding source detection while reducing patient preparation burden compared to standard sequential testing. Results will be compared against conventional approaches to determine optimal diagnostic timing for patients presenting with hematochezia

DETAILED DESCRIPTION:
Gastrointestinal bleeding is a common emergency condition and an important public health issue, as it impacts hospitalization rates and mortality in the population if not properly diagnosed and treated. Currently, GI bleeding is classified into upper GI bleeding, mid GI bleeding, and lower GI bleeding, using the locations accessible by esophagogastroduodenoscopy (EGD) and colonoscopy as the dividing points between the upper, mid and lower GI tracts respectively Patients who present with hematochezia, including passing maroon or bright red blood per rectum, most commonly have lower gastrointestinal bleeding. However, patients with mid or upper gastrointestinal bleeding can also present with hematochezia if bleeding is severe. Thus, colonoscopy is often the first diagnostic test in these patients, able to identify a bleeding source in 68-79% of cases. If no bleeding site is found on colonoscopy, esophagogastroduodenoscopy is then performed, revealing a bleeding lesion in 1.3-15% of patients depending on study population. Those without an identified bleeding site on either colonoscopy or EGD are labeled as potential small bowel bleeders (PSBB). Current guidelines recommend video capsule endoscopy (VCE) in PSBB, since it can detect bleeding sites in 60-70% of these patients.

While the above diagnostic approach is widely accepted, the optimal timing for endoscopic evaluation remains controversial with conflicting study results. Several randomized controlled trials (RCTs) and observational studies have reported higher diagnostic yields and treatment rates when colonoscopy is performed within 24 hours of presentation. Particularly in diverticular bleeding, early colonoscopy enables localization and treatment to prevent rebleeding, since delayed colonoscopy may miss active bleeding once it has spontaneously stopped. However, three RCTs did not show a benefit of urgent colonoscopy. A 2020 meta-analysis also found no improvement in diagnostic yield with urgent colonoscopy in suspected lower GI bleeding. Current guidelines from the American Gastroenterological Association in 2023 also do not recommend urgent colonoscopy. Of note however, in the largest RCT by Niikura et al, the control group underwent colonoscopy at a mean of 41 hours after presentation. The small difference in timing may explain the lack of difference seen between groups.

In addition to timing of colonoscopy, timing of video capsule endoscopy (VCE) also appears to impact diagnostic yields in potential small bowel bleeders. A retrospective cohort study of 94 patients found that urgent VCE within 48 hours of admission increased the diagnosis of small bowel bleeding sources to 66%. A 2022 meta-analysis also showed that early VCE after bleeding increases lesions detection in the small bowel by 4.4-fold.

In summary, urgent colonoscopy does not appear beneficial but urgent VCE increases diagnostic yields in patients presenting with hematochezia. This poses a conflict since urgent VCE necessitates preceding urgent colonoscopy. Thus, this study aims to determine if an approach utilizing urgent colonoscopy within 24 hours followed immediately by same-day VCE in cases of normal colonoscopy can improve bleeding source detection compared to the standard sequential approach. This strategy has not been evaluated before. Additional benefits include reducing bowel preparation requirements for patients. Outcomes will be compared to a group undergoing standard sequential evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admission for maroon stool and/or red blood per rectum with or without hemodynamic instability
3. Hemodynamic stabilization after initial fluid resuscitation
4. Correction of any coagulopathy prior to endoscopy
5. Provision of informed consent

Exclusion Criteria:

1. Hematemesis or nasogastric lavage showing coffee ground material/blood
2. Persistent hemodynamic instability prior to colonoscopy
3. Hospitalization in the preceding 14 days
4. Contraindications to endoscopy e.g. severe asthma, cardiac disease
5. Uncorrected coagulopathy
6. Contraindications to bowel preparation with polyethylene glycol
7. Pregnancy
8. Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of urgent endoscopy compared to standard endoscopy | 72 hour
  The bleeding source detection rate between the urgent endoscopy strategy (colonoscopy + EGD + VCE within 24 hour of presentation) to the standard endoscopy strategy (colonoscopy + EGD + VCE within 72 hour of presentation) will be compared.

SECONDARY OUTCOMES:
Rebleeding rate | 30 days
  The rebleeding rate between the urgent endoscopy strategy group and the standard endoscopy strategy group will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University Bangkok, , Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The investigators are willing to provide our data to researchers who require it. For example, those who want to do systematic review and meta-analysis
Supporting Information: Study Protocol
Time Frame: Other researchers can contact us anytime
Access Criteria: The investigators will provide our protocol and/or data upon request.